CLINICAL TRIAL: NCT05584215
Title: Cognitive Behavioural Therapy-Informed Groups for Psychosis
Acronym: CBTp
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI transitioned to new role
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Serena Wong, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12462
Record Dates: First submitted 2022-06-30; First posted 2022-10-18 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Psychosis
Keywords: cognitive behavioral therapy
MeSH Terms: conditions — Psychotic Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Treatment group will receive cognitive behavioural therapy informed groups for psychosis.
  Interventions: Behavioral: Cognitive Behavioural Therapy for Psychosis Groups
- Control (No Intervention): Control group will be put on a waitlist to receive cognitive behavioural therapy informed groups for psychosis.

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy for Psychosis Groups — Groups based on cognitive behavioural therapy for psychosis
  Arms: Treatment

SUMMARY:
This is a feasibility study of cognitive behavioural therapy-informed groups for psychiatric inpatients with positive symptoms of psychosis.

DETAILED DESCRIPTION:
The majority of inpatients at Parkwood Institute Mental Health have symptoms of psychosis. In line with Health Quality Ontario standards for the treatment of psychosis, the investigators would like to implement and evaluate cognitive behavioural therapy for psychosis (CBTp) informed groups. The feasibility, acceptability, and preliminary efficacy of CBTp groups for inpatients will be examined. Pragmatically, the investigators propose to undergo training in CBTp, implement empirically-supported CBTp protocols developed for inpatients, track outcomes, and publish our findings. The investigators would also incorporate patient feedback to improve future iterations of the protocol. Such an undertaking would build research capacity in front line staff by encouraging engagement in CBTp group training, survey design, participant screening, data collection, analyses, and dissemination of findings.

ELIGIBILITY:
Inclusion Criteria:

* Can read/write in English
* Has positive symptoms of psychosis that are distressing to them

Exclusion Criteria:

* Inability to tolerate group participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-03 (Actual); Primary Completion 2024-01-02 (Estimated); Study Completion 2024-01-02 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcomes in Routine Evaluation 10 (CORE-10) | Up to 2 months
  The Clinical Outcomes in Routine Evaluation 10 is a short 10 item easy-to-use assessment measure for common presentations of psychological distress, designed to be used for screening as well as over the course of treatment to track progress. The minimum value is 0, the maximum value is 40, and higher scores indicate a worse outcome.
Process of Recovery Questionnaire (QPR) | Up to 2 months
  The Process of Recovery Questionnaire is a 15 item questionnaire which was co-produced by people who experience psychosis and their accounts of recovery. The minimum value is 0, the maximum value is 60, and higher scores indicate a better outcome.

SECONDARY OUTCOMES:
The Positive and Negative Syndrome Scale (PANSS) - Positive Symptoms | Up to 2 months
  A brief measure of positive symptoms of psychosis. The minimum value is 7, the maximum values is 49. Higher scores indicate a worse outcome.

OTHER OUTCOMES:
Satisfaction Questionnaire | Up to 2 months
  Brief open-ended questions about program satisfaction. Responses are qualitative.

CONTACTS AND LOCATIONS:
Overall Officials: Serena Wong, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's

IPD SHARING:
Plan to Share IPD: No